CLINICAL TRIAL: NCT03655873
Title: Safety, Tolerability, and Pharmacokinetics Phase ⅠStudy of a Selective 5-ht6 Receptor Antagonist, HEC30654AcOH, Following Single and Multiple Ascending Doses，Single-center, Randomized, Double-blind in Healthy Subjects
Brief Title: The Study of a Selective 5-ht6 Receptor Antagonist, HEC30654AcOH,in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HEC30654-P-01
Record Dates: First submitted 2018-08-24; First posted 2018-08-31 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEC30654AcOH capsule (Experimental): single ascending-dose study: Including 7 dose groups(5-、10、15-、30-、60-、90-、120mg)，Day1 ante meridiem(AM) 8:00 (±1h) with 240ml warm water to taking the experiment drug，On an empty stomach .
  multiple ascending-dose study: Including 3 dose groups(15-、30-、60mg),Day1-Day7 AM 8:00 (±1h), 18:00 Post Meridiem(PM) (±1h), with 240ml warm water to take the experiment drug On an empty stomach;Day8 AM 8:00 (±1h)with 240ml warm water to taking the experiment drug，On an empty stomach.
  Interventions: Drug: HEC30654AcOH capsule
- placebo capsule (Placebo Comparator): single ascending-dose study: Including 6 dose groups(10、15-、30-、60-、90-、120mg)，Day1 morning 8:00 (±1h) with 240ml warm water to taking the placebo capsule，On an empty stomach .
  multiple ascending-dose study: Including 3 dose groups(15-、30-、60mg),Day1-Day7 AM 8:00 (±1h), 18:00 PM (±1h), with 240ml warm water to take the placebo capsule on an empty stomach;Day8 AM 8:00 (±1h)with 240ml warm water to taking the placebo capsule，on an empty stomach.
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: HEC30654AcOH capsule — single ascending-dose study: 5-、10-、15-、30-、60-、90-、120mg HEC30654AcOH capsule in day1.
  Multiple ascending-dose study:
  15-、30-、60mgHEC30654AcOH capsule in day1-day7，2 times everyday.
  Arms: HEC30654AcOH capsule
Drug: Placebo capsule — single ascending-dose study: 5-、10-、15-、30-、60-、90-、120mg placebo capsule in day1.
  Multiple ascending-dose study:
  15-、30-、60mg placebo capsule in day1-day7，2 times everyday.
  Arms: placebo capsule

SUMMARY:
This study is a safety, tolerability, and pharmacokinetics phase Ⅰstudy of a selective 5-ht6 receptor antagonist, HEC30654AcOH,in healthy subjects.This test is divided into two parts, the first part is the healthy adult subjects single ascending-dose research;The second part is the healthy adult subjects multiple ascending-dose research.

DETAILED DESCRIPTION:
The single ascending-dose research:

There have set up seven dose group(5、10、15、30、60、90、120mg）.The first group(5mg)contains 3 health subjects，Which have been a preliminary experimental group. Each other groups contains 10 health subjects(8 health subjects take experimental drugs,2 health subjects take the placebo).Within 15min before taking the medicine and after 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 10h, 12h, 24h, 48h, 72h, 96h, 120h to take blood samples for pharmacokinetics(PK) detection.

The multiple ascending-dose research:

There have set up three dose group(15、30、60mg）.Each group contains 12 health subjects(10 health subjects take experimental drugs,2 health subjects take the placebo).Each dose group in D1-D7 8:00（±1h）in the morning, 18:00（±1h）, with 240 ml warm water to take corresponding study drug，but Day 8 only 8:00（±1h） in the morning take subjects drugs.Total for 15 times.on the morning of day 1 within 15minutes before the first drug and after 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 10h, 12h, on the morning of Day 6, Day 7 and Day 8 within 15 minutes before the drug collecting blood sample test concentration, on the morning of Day8 medication after 0.5h 1h, 1.5h, 2h, 4h, 6h, 8h, 10h, 12h, 24h, 48h, 72h, 96h, 120h collects pharmacokinetics(PK) blood samples.

ELIGIBILITY:
Inclusion Criteria:

* signing informed consent, and fully understanding the study's content, process，possible adverse reaction before the study beginning.
* Be able to complete the study in accordance with the requirements of the study.
* Subjects (including partner) which from screening to the last time of study drug dosage volunteered to take effective contraceptive measures within 6 months, see appendix for birth control measures.
* Age of 18 to 45 years old male and female subjects (including 18 and 45 years of age).
* Male subjects not less than 50 kg, female subjects not less than 45 kg weight.Body mass index (BMI) = weight (kg)/height 2 (m2), body mass index (BMI) within the scope of 18 ~ 28 kg/m2 (including threshold).
* Physical examination, vital signs is normal or abnormal has no clinical significance.

Exclusion Criteria:

* 3 months before the study daily smoking more than 5 pieces.
* having allergies or allergic constitution for experiment drugs (a variety of drugs and food allergies).
* Has a history of drug and/or binge drinking (drinking 14 units of alcohol every week: 1 unit = 285 mL beer, or liquor 25 mL, or wine 100 mL).
* Three months before screening blood or blood loss (> 450 mL).
* 28 days before the screening taking any drugs of changing liver enzymes.
* Within 14 days before the screening taken any prescription drugs, over-the-counter drugs, vitamins or herbal products.
* Within 2 weeks before the screening taking any special diet (including dragon fruit, mango, pomelo, etc.) or with vigorous exercise, or other affect drug absorption, distribution, metabolism and excretion.
* With the following CYP3A4, P - gp or Bcrp inhibitors or inducers, such as itraconazole, ketone health zun or definitely nida, lung, etc.
* Recently, very large changes in diet or exercise habits.
* Three months before taking study drug, there taken study drug and its analogues, or participated in drug clinical trials.
* Having difficulty swallowing or any digestive system diseases history affecting drug absorption, excretion,etc.
* Having had any increased risk of hemorrhagic disease, such as hemorrhoids, acute gastritis or gastric and duodenal ulcer, etc.
* Abnormal ecg that have clinical significance.
* Female subjects in screening test is in lactation or have positive serum pregnancy outcomes.
* Clinical laboratory examination were abnormal clinical significance, or other clinical findings show that there are clinical significance of the following diseases (including but not limited to the gastrointestinal tract, liver, kidney, and nerve, blood, endocrine, tumor, lung, immune, spirit, or disease of heart head blood-vessel).
* Viral hepatitis (including hepatitis b and c),, treponema pallidum antibody , HIV antibody positive.
* From the screening stage to study medicine had a acute disease or taken a drugs.
* Within 48 hours before taking the study drug, there taken any caffeine consumed chocolate, or rich xanthine food or drinks.
* Within 24 hours before taking study drug, there used any alcoholic products or alcohol-breath test was positive.
* Urine drug test(Morphine and marijuana) was positive.
* Neurological examination had abnormal findings, and researchers think have clinical significance.
* Researchers think that doesn't fit to the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events of the single ascending-dose | From the baseline to 6 days
  To assess the safe and tolerability of the single ascending-dose
Adverse events of the multiple ascending-dose | From the baseline to 13 days
  To assess the safe and tolerability of the multiple ascending-dose

SECONDARY OUTCOMES:
Maximum Plasma Concentration(Cmax) | Prior to dosing（0h）and 0.5h,1h,1.5h,2h,4h,6h,8h,10h,12h,24h,48h,72h,96h,120h after dosing
  Maximum Plasma Concentration(Cmax)of HEC30654AcOH in single ascending-dose
Area Under the Curve(AUC) | Prior to dosing（0h）and 0.5h,1h,1.5h,2h,4h,6h,8h,10h,12h,24h,48h,72h,96h,120h after dosing
  Area Under the Curve(AUC) of HEC30654AcOH in single ascending-dose
Maximum Peak Time(Tmax) | Prior to dosing（0h）and 0.5h,1h,1.5h,2h,4h,6h,8h,10h,12h,24h,48h,72h,96h,120h after dosing
  Maximum Peak Time(Tmax) of HEC30654AcOH in single ascending-dose
Mean Residence Time(MRT) | Prior to dosing（0h）and 0.5h,1h,1.5h,2h,4h,6h,8h,10h,12h,24h,48h,72h,96h,120h after dosing
  Mean Residence Time(MRT) of HEC30654AcOH in single ascending-dose
Terminal elimination half-life(T1/2) | Prior to dosing（0h）and 0.5h,1h,1.5h,2h,4h,6h,8h,10h,12h,24h,48h,72h,96h,120h after dosing
  Terminal elimination half-life(T1/2) of HEC30654AcOH in single ascending-dose
steady state plasma concentration(Css） | Prior to dosing（0h）and 0.5h,1h,1.5h,2h,4h,6h,8h,10h,12h after dosing day1,then Prior to dosing（0h）of day6，day7,day8，and 0.5h，1h，1.5h，2h，4h，6h，8h，10h，12h，24h，48h，72h，96h，120h after dosing day8
  steady state plasma concentration(Css）of HEC30654AcOH in multiple ascending-dose

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No